CLINICAL TRIAL: NCT02932475
Title: Medical Optimization of Management of Type 2 Diabetes Complicating Pregnancy
Brief Title: Medical Optimization of Management of Type 2 Diabetes Complicating Pregnancy (MOMPOD)
Acronym: MOMPOD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation by the DSMB that the study be stopped for futility
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-3235; 1R01HD086139-01A1 (NIH)
Record Dates: First submitted 2016-05-17; First posted 2016-10-13 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Pregnancy
Keywords: Metformin; Glucophage; Riomet; Glumetza; Fortamet; Glucophage XR
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Metformin 1000 mg twice a day
  Interventions: Drug: Metformin
- Placebo (Sham Comparator): Placebo, identical to Metformin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 1000 mg twice a day
  Other Names: Glumetza; Fortamet; Glucophage; Riomet
  Arms: Treatment
Drug: Placebo — Delivered to match active drug
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Purpose: The objective of this proposal is to study the safety and efficacy of metformin added to insulin for treatment of type 2 diabetes mellitus (T2DM) among pregnant women.

Participants: 950 pregnant women with type 2 diabetes complicating pregnancy from 10 U.S. clinical centers

Procedures (methods): Pregnant women with T2DM between 10 weeks and 22 weeks 6 days and a singleton fetus will be randomized to double-blinded insulin/placebo versus insulin/metformin. Primary outcome is composite adverse neonatal outcome (clinically relevant hypoglycemia, birth trauma, hyperbilirubinemia, stillbirth/neonatal death). Study visits monthly at clinical visits; blood draw at 24-30 weeks, newborn anthropometric measurements at less than 72 hours of life. Maternal and infant outcomes will be chart abstracted.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18-45 years
* Singleton pregnancy with no known fetal anomalies
* Gestational age between 10weeks 0 days and 22 weeks 6 days by menstrual dating confirmed by ultrasound, or ultrasound alone
* Clinical diagnosis of preexisting T2DM requiring medical treatment (oral agent or insulin)
* Clinical diagnosis of diabetes diagnosed between 10 weeks and < 20 weeks 6 days gestation
* Willing to start insulin therapy and discontinue oral hypoglycemic pills other than study pills
* Able to swallow pills

Exclusion Criteria:

* Clinical diagnosis of pre-existing renal disease, defined as creatinine > 1.5 mg/dL
* Clinical history of lactic acidosis
* Known allergy to metformin
* Participation in another study that could affect primary outcome
* Delivery planned at non-MOMPOD study locations
* Unwillingness to use insulin treatment or follow prenatal care doctor's instructions for insulin and blood glucose monitoring

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 831 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Boggess, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - University of California - San Diego, San Diego, California
  - University of Mississippi, Jackson, Mississippi
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Boggess KA, Valint A, Refuerzo JS, Zork N, Battarbee AN, Eichelberger K, Ramos GA, Olson G, Durnwald C, Landon MB, Aagaard KM, Wallace K, Scifres C, Rosen T, Mulla W, Valent A, Longo S, Young L, Marquis MA, Thomas S, Britt A, Berry D. Metformin Plus Insulin for Preexisting Diabetes or Gestational Diabetes in Early Pregnancy: The MOMPOD Randomized Clinical Trial. JAMA. 2023 Dec 12;330(22):2182-2190. doi: 10.1001/jama.2023.22949. PMID 38085312
- [Derived] Berry DC, Thomas SD, Dorman KF, Ivins AR, de Los Angeles Abreu M, Young L, Boggess K. Rationale, design, and methods for the Medical Optimization and Management of Pregnancies with Overt Type 2 Diabetes (MOMPOD) study. BMC Pregnancy Childbirth. 2018 Dec 12;18(1):488. doi: 10.1186/s12884-018-2108-3. PMID 30541506

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin 1000 mg twice a day
- Placebo: Placebo, identical to Metformin. Delivered to match active drug
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 416 | 415
Randomized | 416 | 415
Received Intervention | 397 | 397
Liveborn Infants During Study | 376 | 370
Completed | 386 | 382
Not Completed | 30 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 397 | 397 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5.5) | 33.1 (5.7) | 32.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 397 | 397 | 794
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 203 | 209 | 412
  Not Hispanic or Latino | 183 | 176 | 359
  Unknown or Not Reported | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 116 | 108 | 224
  White | 55 | 57 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 226 | 232 | 458
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 397 | 397 | 794

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Adverse Neonatal Outcome
Description: Participants with one or more of the following:
  * capillary blood glucose level of < 30 mg/dL or capillary blood glucose requiring medical treatment, or
  * Birth trauma (umbilical cord artery pH < 7.0 or shoulder dystocia with brachial plexus injury), or
  * Hyperbilirubinemia requiring phototherapy, or
  * Deliver < 37 weeks' gestation, or
  * Miscarry, are stillborn, experience a neonatal demise, or
  * Large for gestational age infant (birth weight > 90th percentile for gestational age), or
  * Small for gestational age infant (birth weight < 10th percentile for gestational age) or low birth weight (< 2500 gm)
Time Frame: An average of 48 hours for term infants and 30 days for preterm infants
Population: Modified intent to treat population of all participants who took at least one dose of study agent and had primary outcome data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 386 | 382
Participants | 269 | 277
Statistical Analysis 1: Comparison: Metformin vs Placebo; The sample size gave adequate power over a range of expected primary outcome event rates, with type I error set at 0.044 (reduced from 0.05 for interim analysis), with reasonable power under a conservative scenario assuming that 20% of subjects immediately stopped taking study agent; Test type: Superiority; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.63 to 1.19] — The odds ratio was calculated and adjusted for study site, timing of diabetes diagnosis, gestational age at randomization stratified at 18 weeks, and baseline maternal BMI

2. Secondary Outcome: Number of Participants With Maternal Side Effects
Description: Secondary outcome of maternal side effects were defined as:
  * clinically relevant hypoglycemia defined as capillary blood glucose < 60 or < 80 with symptoms
  * GI side effects defined as nausea, vomiting, diarrhea
Time Frame: Throughout study until delivery at 40 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 397 | 397
Participants
  Clinically relevant hypoglycemia | 87 | 85
  Gastrointestinal side effects | 182 | 171
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.4, Chi-squared — The a priori threshold for statistical significance was <0.05; Difference in proportions = 0.2

3. Secondary Outcome: Mean Infant Fat Mass
Description: Neonatal fat mass measured by skin-fold thickness (anthropometrics).The circumference of the upper limb is the circumference of the upper arm, and the circumference of the lower limb equals the mean of the circumferences measured at the midthigh and calf. The volume of the subcutaneous layer of fat covering each cylinder is estimated by multiplying the length times the circumference times the layer of fat estimated by the skinfold measures. The triceps skinfold measure is used as an estimate of the fat thickness of the limbs, and the subscapular skinfold measure approximates the fat thickness of the trunk. Total body fat is estimated by summing the volumes of fat covering each of the cylinders and multiplying by 0.9 (the density of fat).
Time Frame: Within 72 hrs of birth
Population: Data are reported for those infants who underwent anthropomorphic measurements.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Maternal Metformin: Metformin 1000 mg twice a day
- Maternal Placebo: Placebo, identical to Metformin. Delivered to match active drug
Arm/Group | Maternal Metformin | Maternal Placebo
Number analyzed (Participants) | 218 | 219
kg | 0.46 (0.3) | 0.5 (0.24)
Statistical Analysis 1: Comparison: Maternal Metformin vs Maternal Placebo; Test type: Superiority; p = 0.4, t-test, 2 sided — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = 0.04 — comparison of mean (sd) between groups

4. Secondary Outcome: Maternal Safety Based on Treatment Emergent Adverse Events
Description: Adverse maternal outcomes.
Time Frame: An average of 48 hours following delivery
Population: Number of randomized participants who took at least one dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 397 | 397
Participants
  Any adverse event leading to early study agent discontinuation | 13 | 20
  Any adverse event associated with maternal death | 2 | 1
  Any adverse event associated with fetal death | 10 | 10
  Any maternal serious adverse event | 113 | 111
  Any maternal non-serious adverse event | 149 | 157
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.6, Chi-squared — The a priori threshold for statistical significance is <0.05; Difference in proportions = 0

5. Secondary Outcome: Neonatal Safety Based on Treatment Emergent Adverse Events
Description: Adverse neonatal outcomes
Time Frame: up to 28 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | Maternal Metformin | Maternal Placebo
Number analyzed (Participants) | 376 | 370
Participants
  Any neonatal serious adverse event | 81 | 105
  Any neonatal non-serious adverse event | 157 | 162
Statistical Analysis 1: Comparison: Maternal Metformin vs Maternal Placebo; Test type: Superiority; p = 0.08, Chi-squared — The a priori threshold for statistical significance is <0.05; Difference in proportions = 0

ADVERSE EVENTS:
Time Frame: For mothers, AEs were collected from time of randomization to time of hospital discharge after delivery, an average of 48 hours following delivery. For infants, from birth through 28 days of age.
Groups:
- Fetus of Mother Receiving Metformin: Fetuses in utero to mothers assigned metformin 1000 mg twice a day
- Infants Born to Mothers Receiving Metformin: Infants born to mothers assigned metformin 1000 mg twice a day
- Fetus of Mother Receiving Placebo: Fetuses in utero to mothers assigned placebo delivered to match active drug
- Infants Born to Mothers Receiving Placebo: Infants born to mothers assigned placebo, identical to metformin, delivered to match active drug
Arm/Group | Maternal Metformin | Fetus of Mother Receiving Metformin | Infants Born to Mothers Receiving Metformin | Maternal Placebo | Fetus of Mother Receiving Placebo | Infants Born to Mothers Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 2/397 | 10/397 | 1/376 | 1/397 | 10/397 | 2/370
Serious Adverse Events (participants affected / at risk) | 113/397 | 0/397 | 81/376 | 111/397 | 0/397 | 105/370
Other Adverse Events (participants affected / at risk) | 54/397 | 0/397 | 151/376 | 57/397 | 0/397 | 151/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Metformin (N=397) | Fetus of Mother Receiving Metformin (N=397) | Infants Born to Mothers Receiving Metformin (N=376) | Maternal Placebo (N=397) | Fetus of Mother Receiving Placebo (N=397) | Infants Born to Mothers Receiving Placebo (N=370)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain' (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperemesis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HELLP Syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Asthma (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Postop wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postop wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 8 (8) | 2 (2) | 0 (0) | 13 (13)
Gastroparesis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 44 (44) | 0 (0) | 0 (0) | 32 (32) | 0 (0) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Preterm labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 19 (19) | 2 (2) | 0 (0) | 22 (22)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puerperal infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shortened cervix (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Social circumstances (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Homeless (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix cerclage procedure (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placental insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Persistent foetal circulation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Truncus arteriosus persistent (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal atresia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Beckwith-Wiedemann syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 9 (9)
Pulmonary malformation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sequestration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal testicular torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genitalia external ambiguous (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infantile apnoea (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Immature respiratory system (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 8 (8)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 19 (19) | 0 (0) | 0 (0) | 22 (22)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Metformin (N=397) | Fetus of Mother Receiving Metformin (N=397) | Infants Born to Mothers Receiving Metformin (N=376) | Maternal Placebo (N=397) | Fetus of Mother Receiving Placebo (N=397) | Infants Born to Mothers Receiving Placebo (N=370)
Abdominal pain (Gastrointestinal disorders) | 23 (23) | 0 (0) | 0 (0) | 20 (20) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 31 (31) | 0 (0) | 0 (0) | 36 (36) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 56 (56) | 1 (1) | 0 (0) | 54 (54)
Jaundice (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 95 (95) | 0 (0) | 0 (0) | 97 (97)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02932475/Prot_SAP_000.pdf